

Title: A 3-Part, Randomized, Double-Blind, Placebo-Controlled, Multiple Rising Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TAK-925 in Healthy Volunteers and Patients with Narcolepsy

NCT Number: NCT03748979

Statistical analysis plan Approve Date: 28-OCT-2019

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).



A 3-Part, Randomized, Double-Blind, Placebo-Controlled, Multiple Rising Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TAK-925 in Healthy Volunteers and Patients with Narcolepsy

Version: 2<sup>nd</sup>

Date: 28 October 2019 AK-925
acebo-Controlled,
narmacokinetics and P.
anteers and Patients with N

Version: 2<sup>nd</sup>

Date: 28 October 2019

Date: 28 October 2019

Ny:

Prepared by:

PPD

Based on:

Protocol Version: Amendment 3

Property of Lakedai. Protocol Date: 12 June 2019

Properly of Takeda, for nonconfine cial use only and subject to the applicable Terms of Use

## 2.0 TABLE OF CONTENTS

| | 1.1 | CCI | | 2 |
|---|---|---|---|---|
| 2.0 | | | E OF CONTENTS | |
| 3.0 | | LIST ( | OF ABBREVIATIONS | 5 |
| 4.0 | | TRIAI | L OBJECTIVES | X |
| | 4.1 | Tri | ial Primary Objectives | |
| | 4.2 | Tri | ial Secondary Objectives | 7 |
| | 4.3 | Tri | ial Exploratory Objectives | <i>7</i> |
| | 4.4 | Tri | ial Secondary Objectives ial Exploratory Objectives ial Design | 8 |
| 5.0 | | ANAL | Primary Endpoint Secondary Endpoints | 12 |
| | | 5.1.1 | Primary Endpoint | 12 |
| | | 5.1.2 | Secondary Endpoints | 12 |
| | | 5.1.3 | CCI | 12 |
| | | 5.1.4 | CCI | 12 |
| 6.0 | | | RMINATION OF SAMPLE SIZE | |
| 7.0 | | | HODS OF ANALYSIS AND PRESENTATION | |
| | 7.1 | Ge | Study Definitions | 15 |
| | | 7.1.1 | Study Definitions | 15 |
| | 7.2 | An | nalysis Sets | 16 |
| | 7.3 | Dis | sposition of Subjects Study Information | 17 |
| | | 7.3.1 | Study Information | 17 |
| | | 7.3.2 | Screen Failures. | 17 |
| | | 7.3.3 | Subject Eligibility | |
| | | 7.3.4 | Disposition of Subjects | |
| | | 7.3.5 | Protocol Deviations and Analysis Sets | |
| | 7.4 | | emographic and Other Baseline Characteristics | |
| | | X | Cohort A1~A3 | |
| | | 7.4.2 | Cohort B1~B2 | 23 |
| | V | 3.4.3 | Cohort C1~C2 | |
| < | <u>ر</u> ، | 7.4.4 | Cohort A'1 | |
| | 7.5 | | edical History and Concurrent Medical Conditions | |
| | | 7.5.1 | Cohort B1~B2 | |
| | 7.6 | 7.5.2 | Cohort C1~C2 | |
| | 7.6 | 7.6.1 | edication History and Concomitant Medications | |
| | | , | | |
| | 7.7 | | Cohort C1~C2 | |
| | /./ | | ady Drug Exposure and Compliance | 20 |

| Statistical Linux | , 515 1 IMI 2110 | TO OTTOBER TO |
|---|---|---|
| 7.7.2 | Cohort B1~B2 | 26 |
| 7.7.3 | Cohort C1~C2 | |
| | ficacy Analysis | |
| 7.8.1 | Primary Efficacy Endpoint(s) | |
| 7.8.2 | Secondary Efficacy Endpoint(s) | |
| 7.8.3 | Additional Efficacy Endpoint(s) | |
| 7.8.4 | Statistical/Analytical Issues | 37 |
| | armacokinetic/Pharmacodynamic Analysis | |
| 7.9.1 | Pharmacokinetic Analysis | 28 |
| 7.9.2 | Pharmacokinetic Analysis Pharmacodynamic Analysis | 32 |
| 7.10 | | 40 |
| 7.10.1 | CCI | |
| | | 40 |
| 7.11 Sa | fety Analysis Adverse Events Clinical Laboratory Evaluations | 43 |
| 7.11.1 | Adverse Events | 43 |
| 7.11.2 | Clinical Laboratory Evaluations | 48 |
| 7.11.3 | | 51 |
| 7.11.4 | CCI | 54 |
| 7.11.5 | CCI | 56 |
| 7.11.6 | CCI | 57 |
| 7.11.7 | CCI | 58 |
| 7.11.8 | Other Observations Related to Safety | 58 |
| | erim Data Review | |
| | nanges in the Statistical Analysis Plan | 58 |
| | EFERENCES | |
| APPENDIX A | A CCI | |
| | | 82 |
| < | 0, | |
| LICT OF DE | TEVT TADI EC | |

# LIST OF IN-TEXT TABLES

### LIST OF ABBREVIATIONS 3.0

ΑE

ALT ANCOVA AST

**AUC** 

BMI BP

Ceoi CL

Cmax

andex

and pressure

plasma concentration at the end of infusion

total clearance after intravenous administration

maximum observed concentration

coefficient of variation

lectrocardiogram

'ectroencephalography

worth sleeping

mma-c' CV**ECG EEG** ESS GGT gamma-glutamyl transferase Good Clinical Practice **GCP** healthy volunteer HV

Independent Ethics Committee **IEC** Institutional Review Board **IRB** 

intravenous IV

karolinska sleepiness scale **KSS** dactate dehydrogenase LDH

LS least square

MAV markedly abnormal value mean cell hemoglobin **MCH** 

**MCHC** mean cell hemoglobin concentration

MCV mean cell volume

MedDRA medical dictionary for regulatory activities

MR metabolic ratio MRD multiple rising dose

**MWT** maintenance of wakefulness test

narcolepsy type 1 NT1 NT2 narcolepsy type 2 PD pharmacodynamics

PGI-C patient global impression of change

pharmacokinetics PK

PT preferred term PTE pretreatment event

**PTR** peak trough ratio during a dosing interval, at steady state

**PVT** psychomotor vigilance task

QT interval corrected for heart rate by the Bazett method **QTcB** QT interval corrected for heart rate by the Fridericia method **QTcF** 

**RBC** red blood cell

accumulation ratio based on AUC during a dosing interval Rac AUC

Rac Cmax accumulation ratio based on Cmax and subject

**REM** rapid eye movement

reaction time RT

serious adverse event SAE statistical analysis plan SAP SD standard deviation SOC system organ class

treatment-emergent adverse event **TEAE** time of first occurrence of Cmax tmax

half-life period t1/2z

volume of distribution at state after intravenous administration Vss

volume of distribution VzProperty of Lakedai. For hon.c white blood cell

World Health Organization Drug Dictionary

### 4.0 TRIAL OBJECTIVES

To investigate the safety and tolerability of TAK-925 when administered to healthy subjects and NT1 and NT2 patients.

4.2 Trial Secondary Objectives

<All parts>

To investigate the pharmacokinetics of TAK-925 when administered to healthy volunteers or narcolepsy patients

<Part B and C>

To investigate the PD of TAK-925 after multiple doses, primarily with evaluation of sleep latency on MWT when TAK-925 is administered to NT1 and NT2 patients.

4.3 **Trial Exploratory Objectives** 





## 4.4 Trial Design

This study will consist of 3 parts. Part A is a randomized, double-blind, placebo-controlled, MRD study to assess safety, tolerability, and PK of TAK-925 administered via intravenous (IV) infusion in healthy subjects. Part B is a randomized, double-blind, placebo-controlled MRD study to assess the safety, tolerability, PK and PD of TAK-925 administered via IV infusion in patients with NT1. Part C is a randomized, double-blind, placebo-controlled, parallel group multiple repeat dose study to assess the safety, tolerability, PK and PD of one or more dose levels of TAK-925 vs. placebo in patients with NT2. Part A' is an open-label single oral dose study to assess PK, safety and tolerability of TAK-925 administered orally in healthy subjects. Parts A - A' may be conducted in parallel, rather than sequentially, depending on the doses administered and emerging safety/tolerability data.

In general, considering the completion times of the prior studies, TAK-925-1001 and TAK-925-1002, Part A, Part B and Part A' are expected to begin in parallel. Part A will test safety and tolerability in healthy volunteers (HV) starting from the dose level associated with that was found to be safe and tolerable based on the preliminary blinded safety adverse event (AE) profiles in TAK-925-1001 study. Part B will test safety, tolerability and PD in NT1 patients, who will be administered a lower dose than subjects in Part A. The initial dose in Part B was found to be safe and tolerable based on the preliminary blinded safety AE profiles in NT1 patients in the TAK-925-1001 study. The initial dose in Part B is more than 10 times lower than the highest dose level tested in TAK-925-1001 HV cohorts. Results from the TAK-925-1001 study will also be available at the time of initiation of Part A and Part B. Part A' will assess the safety, tolerability and CC TAK-925 to healthy volunteers at a dose level that was found to be safe and tolerable after IV administration in TAK-925-1001 study and is anticipated to result in lower exposure of TAK-925 after oral administration,

For Part C, the NT2 patient doses are expected to be similar to that in Part A, although recruitment of these cohorts will be slower. Initiation of Part A and Part C may also occur at the same time if the similar doses are studied. The initiation of cohorts in parallel with each other is contingent on Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approval, and if not approved, the cohorts will enroll as required, which may be sequentially or overlapping with each other. The NT1 and NT2 patients recruited are expected to be generally healthy other than having narcolepsy.

Part A will have 2 dose cohorts as well as additional 4 optional cohorts. Each cohort of healthy adults will consist of 8 healthy subjects, randomized 6:2 active to placebo to TAK-925 vs. placebo (Table 4.a) in double-blinded fashion. The starting dose is selected based on the available preliminary safety, PK and PD data from the ongoing TAK-925-1001 study. Subsequent doses will be guided by safety, PK and PD data from previous cohorts as well as the TAK-925-1002 study (which is ongoing at the time of this protocol writing). TAK-925 or placebo will be administered as an IV infusion over 9 hours once daily for 7 days. Following review of emerging safety and PK data (when available) in Cohort A1, the dose in Cohort A2 will be determined. Healthy adults may be recruited for up to 3 additional cohorts (A3 to A5) with 8 subjects each (randomized 6:2 active to placebo). The dose may be higher, lower or the same as that of prior cohort dose levels. Shifting the start time of infusion while keeping the dose the same as that previously studied may be considered in these optional cohorts . The maximum dose and infusion rate in Part A shall not exceed the maximum dose or maximum infusion rate studied in healthy subjects in TAK-925-1001 study. The dose levels in subsequent cohorts will be optimized based on the recommendation of sponsor's unblinded team. The unblinded team will review available unblinded data including

The safety and tolerability of the same or a lower dose than that of previous healthy adults cohorts may be studied in an optional cohort of healthy elderly subjects (N=8 subjects aged 65-80 years old, randomized 6:2 to TAK-925 vs. placebo) in Cohort A6. The healthy elderly optional cohort will be included as there are expected to be a few older patients in the Part B or Part C. It is expected that the healthy elderly cohort will provide data that supports the evaluation of TAK-925 in

### Part B – Multiple Rising Dose in Narcolepsy Type 1 (NT1) Patients

Part B will be conducted in NT1 patients. Two cohorts are planned, with optional cohorts allowed. For Cohorts B1 and B2, each cohort will consist of 6 subjects, randomized 4:2 to TAK-925 vs. placebo (Table 4.a) in double blinded fashion. TAK-925 or placebo will be administered as an IV infusion over 9 hours once daily for 7 days. Exploratory PD assessments will include evaluation of potential efficacy with

The starting dose level in Part B will be selected based on preliminary data from the ongoing TAK-925-1001 study utilizing data regarding safety and tolerability, PK and results on the KSS and MWT in the NT1 cohorts, as well as the safety, tolerability and PK results in the healthy adult cohorts in TAK-925-1001 and Part A of this study (if available). The doses in the subsequent cohorts will be determined based on safety, tolerability, PD and available PK data from previous cohorts and/or from the prior studies with TAK-925. The dose level chosen in each of the subsequent cohorts will be determined by the sponsor's unblinded team composed of personnel who do not have subject contact or involvement with execution of the protocol at the site. The unblinded team will review unblinded safety, tolerability, and available PK and PD results from previous cohorts. The dose in the subsequent cohorts may be higher, the same as or lower than that used in the previous cohort(s).

Two additional cohorts (B3 and B4) may be evaluated, with 4-6 subjects in each. With the intention of sequential panel design, NT1 patients in Cohort B1 or B2 may participate in Cohort B3 or B4 if feasible operationally. Patients in cohort B1 and B2 may participate in B3 or B4 after a sufficient washout period if and allowed by regulatory authorities and IRB/IEC. The subject who directly move on to cohort B3 or B4 could skip the Day 8 some assessments and follow up visit and move into Day-2 in B3 or B4. Cohort B3 or B4 will essentially consist of newly enrolled NT1 patients, but patients from B1/B2 who weigh over 50 kg could be also enrolled. There should be sufficient intervals between the last dose in Cohort B1 or B2 and the first dose in Cohort B3 or B4 in order to make dose and dosing duration decisions for Cohorts B3 and B4. If there are fewer than 4 Cohort B1 or B2 subjects enrolled to Cohort B3 or B4, new patients with NT1 will be recruited. In Cohorts B3 and B4, TAK-925 will be administered in a blinded randomized manner (3:1, 4:1 or 5:1). The primary purpose of Cohort B3 is to evaluate the safety and tolerability and PD of longer infusion time, as well as to

Otherwise, the design and procedures for B3 will be the same as the design of B1. The primary purpose of Cohort B4 is to assess the within-subject exposure-response relationship for PD/efficacy and safety of TAK-925 in NT1 patients. Patients in this cohort will receive different, increasing doses of TAK-925 daily over the 7 day period, the sequence of doses will be identical across patients. All subjects will receive the same dosing schedule. One subject within B3 and B4, respectively, will be randomized to placebo.

## Part C – Multiple Doses in Narcolepsy Type 2 (NT2) patients

Narcolepsy type 2 patients will be evaluated in Cohorts C1 and C2. This part will start once TAK-925-1002 study data is available and once safety/tolerability information for the dose level to be tested in Part C is available from Part A. Conduct of the C2 cohort is optional. C1 and C2 cohorts will recruit 6 subjects each, randomized 4:2 to TAK-925 vs. placebo in double-blinded fashion, with study drug administered as a 9-hour intravenous infusion for 7 days (Table 4.a). The doses selected for Part C depend on the results from the TAK-925-1002 study, and data from other cohorts in this study may also be used. The same schedule of study assessments as in Part B will be executed

### Part A' - Single Oral Doses in Healthy Adults

Part A' will investigate the pharmacokinetics of TAK-925 after oral administration in healthy subjects. Cohort A'1 will consist of 6 healthy subjects who will be administered a single dose of TAK-925 as an oral solution in an open-label fashion (Table 4.a). An oral dose of 112 mg is selected based on the safety and tolerability profiles in TAK-925-1001 study and available nonclinical data as a potential starting dose.

925- An optional Cohort A'2 is allowed based on the emerging information.

The study parts and planned dosing cohorts are outlined in Table 4.a.

**Outline of the Study Parts and Planned Dosing Cohorts** Table 4.a

| Part | Cohort/Panel | Daily dose level (mg) | Dosing regimen | Randomization |
|---|---|---|---|---|
| | A1 | 44 | | 8 subjects randomized 6:2 to TAK-925 vs. placebo in each cohort, double-blind 6 subjects randomized 4: 2 to TAK-925 vs. placebo in each cohort, double blind |
| | A2 | 112 (TBD) | IV infusion over 9 hours | |
| Part A | A3* | TBD | up to 7 days. Start time of infusion could be changed | |
| (Healthy adults)# | A4* | TBD | in optional cohorts A3 to | |
| | A5* | TBD | A5. | |
| | A6 (elderly)* | TBD | ] | |
| | B1 | 11 | | |
| | B2 | 44 (TBD) | IV infusion over 9 hours up to 7 days | |
| Part B (NT1 patients)# | B3* | TBD | IV infusion with longer (TBD) hours up to 7 days | 4-6 subjects randomized |
| | B4* | TBD | IV infusion over 9 hours<br>up to 7 days, different,<br>increasing dose from Day<br>1 to Day 7 | (3:1, 4:1 or 5:1 to TAK-<br>925 vs. placebo in each<br>cohort, double blind |
| | C1 | 44 (TBD) | and | 6 subjects randomized 4: |
| Part C (NT2 patients)# | C2* | TBD ON | W infusion over 9 hours<br>up to 7 days | 2 to TAK-925 vs. placebo<br>in each cohort, double<br>blind |
| Part A' (Healthy | A'1 | 112 | | |
| adults) | A'2* | TBD | Single oral administration | (TAK-925 administration, open) |

Doses in subsequent cohorts in all parts will be determined based on the emerging safety/tolerability and PK (when available) and PD information and available safety/tolerability, and PK/PD data from previous cohorts as well as the ongoing TAK-925-1001 and TAK-925-1002 studies. Planned number of subjects in each cohort is Property of Pakeda.

<sup>#</sup> All doses given by IV infusion over 9 hours daily for 7 days except B3

### 5.0

### 5.1.1 Primary Endpoint

<All Parts>

• Safety and tolerability: number of subjects with AEs

## **5.1.2** Secondary Endpoints

< Parts A, B and C>

• Pharmacokinetic parameters ( $C_{eoi}$ , AUC  $_{\tau}$ ,  $R_{ac(AUC)}$ ) of TAK-925

<Part B and C>

5.1.4

JOKINETIC parameters (Ceoi, AUC, Rac(AUC)) of TAK-925

Yart B and C>

Change from baseline in Sleep latency in the MWT to Days 1 and Recommendations of the state 5.1.3

.AMPLE SIZE

.ojects per cohort: 6 active and 2 placebo), Part 1.
and 2 placebo) and Part A' (open label, 6 subjects per or investigating the safety, tolerability, pharmacokinetics, iAK-925 when multiple does of TAK-925 are administered athy adults, healthy elderly, and narcolepsy patients, or when a sin, is administered orally in healthy adults. The sample size is not based to of statistical power. placebo), Part B and C (6 per label, 6 subjects per cohort) is part and pharmacodynamics of TAK-925 when multiple doses of TAK-925 are administered intravenously in healthy adults, healthy elderly, and narcolepsy patients, or when a single dose of TAK-925 is administered orally in healthy adults. The sample size is not based on considerations of statistical power.

### 7.0 METHODS OF ANALYSIS AND PRESENTATION

## 7.1 General Principles

## 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- Treatment-emergent adverse event (TEAE): An adverse event that occurs on or after the start of study drug administration.
- Pretreatment event (PTE): Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to administration of study drug
- Descriptive statistics: Number of subjects, mean, standard deviation, maximum, minimum, and quartiles
- Coefficient of variation (CV) (%): Standard deviation / mean \* 100
- Average Sleep Latency in MWT: Average of four MWTs measured on the same day
- QTcF interval (msec): QT interval (msec) / (RR interval (sec))<sup>0.33</sup> (rounded to the nearest whole number)
- Period for diagnosis (year): The value of age of onset subtracted from the value of age at date of informed consent
- Change from time-matched baseline: Values of Day -1 subtracted from values of Day 1 and 7 in the matching column in the table below for each subject

| K | | TT T | _ |
|---|------|-----------|---|
| | N /I | \ \ \ / · | |
| | 11/1 | VV | |

| Day | Time (Time postdose (hour) ) | | | |
|---|---|---|---|---|
| Day -1 | 10:00 | 12:00 | 14:00 | 16:00 |
| Day 1,7 | 10:00 (2 hr) | 12:00 (4 hr) | 14:00 (6 hr) | 16:00 (8 hr) |





- Time-matched baseline: observed value of Day -1 obtained time-matched with Day1 and 7 in the table above for each subject
- Change from Time-matched Day 1 to Day 7: For MWT and vital sign parameters, values
  of Day 1 subtracted from values of Day 7 in the matching column in the table above for
  each subject
- Treatment Group
  - Cohort A1~A3
    - ♦ Placebo (pooled Cohort A1, A2 and A3)
    - ♦ TAK-925 44mg, 112mg, 180mg
  - Cohort B1~B2
    - ♦ Placebo (pooled Cohort B1 and B2)
    - ♦ TAK-925 11mg, 44mg
  - Cohort C1~C2
    - ♦ Placebo
    - ♦ TAK-925 44mg, 112mg
  - Cohort A'1
    - \*TAK-925 112mg

### 7.2 Analysis Sets

- Safety set: All subjects who received at least one dose of study drug
- PK set: All subjects who received at least one dose of study drug and provided sufficient PK measurements available to estimate PK parameters, at least 1 estimable PK parameter.
- PD set: All subjects who received at least one dose of study drug.

### 7.3 **Disposition of Subjects**

### 7.3.1 **Study Information**

All Subjects Who Signed the Informed Consent Form Analysis Set:

Analysis

Variable(s): Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version

SAS Version Used for Creating the Datasets

Analytical

Method(s): (1) Study Information

the applicable terms of Use ion Study information shown in the analysis variables section will be provided.

### 7.3.2 **Screen Failures**

All Subjects Who Were Not Randomized Analysis Set:

Analysis

Variable(s): Age (years)

> [Male, Female] Gender

Analytical

(1) Screen Failures Method(s):

Frequency distributions for categorical variables and descriptive statistics

for continuous variables will be provided.

### **Subject Eligibility**

## 7.3.3.1 Cohort A1~A3

nalysis Variable(s): Analysis Set: All Subjects Who Signed the Informed Consent Form

Study Drug Administration Status

Primary Reason for Subject Not

Being Treated

[Rnadomized, Not Randomized]

[Adverse Event, Death, Lost to

Follow-up, Pregnancy, Protocol

Deviation, Sample Size Sufficient,

Screen Failure, Study Terminated by

Sponsor, Withdrawal by Subject,

Other]

Analytical

Method(s): (1) Study Drug Administration Status

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being treated, the total number of not treated subjects will be used as the denominator.

7.3.3.2 Cohort B1~B2

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analytical

Method(s): The same analysis as section 7.3.3.1 will be performed for the Cohort

B1~B2

7.3.3.3 Cohort C1~C2

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analytical

Method(s): The same analysis as section 7.3.3.1 will be performed for the Cohort

C1~C2

7.3.3.4 Cohort A'1

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analytical

Method(s): The same analysis as section 7.3.3.1 will be performed for the Cohort A'1

7.3.4 Disposition of Subjects

7.3.4.1 **C**ohort A1~A3

Analysis Set: All Subjects Who Received Study Drug

Analysis

Variable(s): Study Completion Status [Completed All Planned Study

Visits, Did Not Complete All

Planned Study Visits]

Reason for Discontinuation of

Study Visits

[Adverse Event, Death, Lost to Follow-up, Pregnancy, Protocol

Deviation, Study Terminated by

Sponsor, Withdrawal by Subject, Other]

Analytical

Method(s): (1) Disposition of Subjects

Frequency distributions will be provided by treatment group and overall. When calculating percentages for the reasons for discontinuation, the total number of subjects who did not complete all planned study visits will be used as the denominator.

### 7.3.4.2 Cohort B1~B2

Analysis All Subjects Who Received Study Drug

Set:

Analytical

Method(s): The same analysis as section 7.3.4.1 will be performed for the Cohort  $B1\sim B2$ 

### 7.3.4.3 Cohort C1~C2

Analysis All Subjects Who Received Study Drug

Set:

Analytical

Method(s): The same analysis as section 7.3.4.1 will be performed for the Cohort C1~C2

### 7 3 4 4 Cohort A'1

Analysis Set: All Subjects Who Received Study Drug

Analytical .

Method(s): The same analysis as section 7.3.4.1 will be performed for the Cohort A'1

## 7.3.5 Protocol Deviations and Analysis Sets

### 7.3.5.1 Protocol Deviations

### Cohort A1~A3

Analysis Set: All Subjects Who Received Study Drug

Analysis

Variable(s): Significant Protocol

Deviation

reims of Use [Entry Criteria, Concomitant Medication, Procedure Not Performed Per Protocol, Study Medication, Withdrawal Criteria, Major GCP Violations]

Analytical

Method(s): (1) Protocol Deviations

> Frequency distribution will be provided by treatment group and overall for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

### Cohort B1~B2

All Subjects Who Received Study Drug Analysis

Set:

Analytical

The same analysis as section 7.3.5.1 "Cohort A1~A3" will be performed for Method(s):

the Cohort B1~B2

### Cohort C1~C2

All Subjects Who Received Study Drug Analysis

Set:

The same analysis the Cohort C1~C2 The same analysis as section 7.3.5.1 "Cohort A1~A3" will be performed for

### Cohort A'1

Analysis Set:

Analytical

The same analysis as section 7.3.5.1 "Cohort A1~A3" will be performed for the Cohort A'1

s Sets

All Subjects Who Received Study Drug

Handling of Subjects Method(s):

## 7.3.5.2 Analysis Sets

### Cohort A1~A3

Analysis Set: All Subjects Who Received Study Drug

Analysis

Variable(s):

specifications in Subject Evaluability

List]

Analysis Sets

Safety Set [Included] PK Set [Included]

Analytical

(1) Subjects Excluded from Analysis Sets Method(s):

(2) Analysis Sets

Frequency distributions will be provided by treatment group and overall. For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

All Subjects Who Received Study Drug

Analysis

Variable(s): Handling of Subjects [Categories are based on the

specifications in Subject Evaluability

List]

Analysis Sets

Safety Set [Included] PK Set [Included]
PD Set [Included]

Analytical

Method(s): The same analysis as section 7.3.5.2 "Cohort A1~A3" will be performed for

the Cohort B1~B2

### Cohort C1~C2

Analysis All Subjects Who Received Study Drug

Set:

Analysis

Variable(s): Handling of Subjects [Categories are based on the

specifications in Subject Evaluability

List]

Analysis Sets

Safety Set [Included]
PK Set [Included]
PD Set [Included]

Analytical

Method(s): The same analysis as section 7.3.5.2 "Cohort A1~A3" will be performed for

the Cohort C1~C2

### Cohort A'1

Analysis Set: All Subjects Who Received Study Drug

Analytical

Method(s): The same analysis as section 7.3.5.2 "Cohort A1~A3" will be performed for

the Cohort A'1

# 7.4 Demographic and Other Baseline Characteristics

### 7.4.1 Cohort A1~A3

Analysis Set: Safety Set

Analysis

Variable(s): Age (years)

Gender [Male, Female]

Height (cm)

Weight (kg)

BMI  $(kg/m^2)$ 

Analytical

Method(s):

(1) Summary of Demographics and Baseline Characteristics Frequency distributions for categorical variables and descriptive statistics and subject to for continuous variables will be provided by treatment group and overall.

## 7.4.2 Cohort B1~B2

Analysis Set: Safety Set

Analysis

Variable(s): Age (years)

Gender

Height (cm)

Weight (kg)

BMI  $(kg/m^2)$ 

 $[Min \le - <65, 65 \le - <=Max]$ 

[Never, Current, Former]

[Daily, A Few Times Per Week, A

Few Times Per Month, No]

[Yes, No]



Age of onset (year)

Period for diagnosis (year)



Analytical

(1) Summary of Demographics and Baseline Characteristics Method(s):

icable Terms of Use Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided by treatment group and overall.

### 7.4.3 Cohort C1~C2

Analysis Set: Safety Set

Analytical

The same analysis as section 7.4.2 will be performed for the Cohort C1~C2 Method(s):

### 7.4.4 Cohort A'1

Analysis Set: Safety Set

Analytical

The same analysis as section 7.4.1 will be performed for the Cohort A'1 Method(s):

### 7.5 **Medical History and Concurrent Medical Conditions**

### Cohort B1~B2 7.5.1

Analysis Set: Safety Set

Analysis

Variable(s): Medical History

**Concurrent Medical Conditions** 

Analytical

Method(s): (1) Medical History by System Organ Class and Preferred Term

> (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided for each treatment group and overall. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and

Exercences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

C1~C2

Safet

### 7.5.2 Cohort C1~C2

Analysis Set: Safety Set

Analytical

The same analysis as section 7.5.1 will be performed for the Cohort C1~C2 Method(s):

### **Medication History and Concomitant Medications** 7.6

### Cohort B1~B2 7.6.1

Analysis Set: Safety Set

Analysis

Variable(s): **Medication History** 

Concomitant Medications

Analytical

Method(s): (1) Medication History by Preferred Medication Name

- (2) Concomitant Medications That Started and Stopped Prior to Baseline by Preferred Medication Name
- (3) Concomitant Medications That Started Prior to and Were Ongoing at Baseline by Preferred Medication Name
- (4) Concomitant Medications That Started After Baseline by Preferred Medication Name
  - (5) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by Preferred Medication Name

Frequency distributions will be provided for each treatment group and overall. A summary of (2)  $\sim$  (5) will also be provided for concomitant medications whose primary purpose was "primary diagnosis". WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several

medications with the same preferred medication name will be counted only once for that preferred medication name.

### 7.6.2 Cohort C1~C2

Analysis Set: Safety Set

Analytical

The same analysis as section 7.6.1 will be performed for the Cohort C1~C2 Method(s):

### 7.7 **Study Drug Exposure and Compliance**

### 7.7.1 Cohort A1~A3

Analysis Set: Safety Set

Analysis

[1, 2, 3, 4, 5, 6, 7] Number of Times the Study Drug was Taken Variable(s):

Analytical

(1) Study Drug Exposure Method(s):

Frequency distributions will be provided by treatment group.

### Cohort B1~B2 7.7.2

Analysis Set: Safety Set

Analytical

The same analysis as section 7.7.1 will be performed for the Cohort B1~B2 Method(s):

### 7.7.3 Cohort C1~

Analysis Set: Safety Set

Analytical

Method(s): The same analysis as section 7.7.1 will be performed for the Cohort C1~C2

## **Efficacy Analysis**

Not applicable.

### 7.8.1 Primary Efficacy Endpoint(s)

Not applicable.

### 7.8.2 Secondary Efficacy Endpoint(s)

Not applicable.

## 7.8.3 Additional Efficacy Endpoint(s)

Not applicable.

### 7.8.4 Statistical/Analytical Issues

7.8.4.1 Adjustments for Covariates

Not applicable.

7.8.4.2 Handling of Dropouts or Missing Data

No imputations will be performed for missing PD (exclude ) and safety measures.

-Jable reinis of Use

For plasma concentrations and laboratory test results, values below the lower limit of quantification will be treated as zero when calculating the descriptive statistics.

only and subje

7.8.4.3 Multicenter Studies

Not applicable.

7.8.4.4 Multiple Comparison/Multiplicity

Not applicable.

7.8.4.5 Use of an "Efficacy Subset" of Subjects

Not applicable.

7.8.4.6 Active-Control Studies Intended to Show Equivalence or Non-Inferiority

Not applicable.

7.8.4.7 Examination of Subgroups

Not applicable of the desired of the

- Pharmacokinetic/Pharmacodynamic Analysis 7.9
- 7.9.1 Pharmacokinetic Analysis

7.9.1.1





Property



Property of Lakeda.

## 7.9.1.2 Pharmacokinetic Parameters

### Cohort A1~A3

Analysis Set: PK Set

Analysis

Variable(s): Pharmacokinetic Parameters of TAK-925 and



Visit:

Day 1, Day 7

Analytical

The following summaries will be provided by treatment group. Subjects Method(s): administered placebo will be excluded from the analysis.

> (1) Summary of Pharmacokinetic Parameters , AUCtau, Ceoi, descriptive

statistics, geometric mean, and CV will be provided.

(2)

# Cohort B1

Analysis Set: PK Set

Analytical

Method(s): The same analysis as section 7.9.1.2 "Cohort A1~A3" will be conducted for

the Cohort B1~B2.

## Cohort C1~C2

Analysis Set: PK Set

Analytical

The same analysis as section 7.9.1.2 "Cohort A1~A3" will be conducted for Method(s):

the Cohort C1~C2.





# Pharmacodynamic Analysis

Average Sleep Latency in MWT/Sleep Latency in Each Session in MWT

## Cohort B1~B2

Analysis Set: PD Set

Analysis

√aria Visit: Variable(s): Average Sleep Latency in MWT, Sleep Latency in Each Session in MWT

Average Sleep Latency in MWT: Day -1, Day 1, Day 7

Sleep Latency in Each Session in MWT:

Day -1: 10: 00, 12: 00, 14: 00, 16: 00

Day 1 and Day 7: 10:00 (2hr), 12:00 (4hr), 14:00 (6hr), 16:00 (8hr)

Analytical

Method(s): The following summaries will be provided.

(1) For the average sleep latency in MWT, descriptive statistics for the

, changes from baseline and

treatment of TAK-925 and placebo), day (as a categorical variable), the treatment-by-day as fixed effects, baseline average sleep latency in the MWT as a covariate, and subjects as a randomeans, the standard will be provided by visit by treatment group. The effect of TAK-925 will be provided for each treatment group. For each day, the difference in the LS means between each treatment of TAK-925 and the placebo (each treatment of TAK-925 - the placebo), the standard error of the difference and the two-sided confidence intervals will be provided.

The differences in the LS means between each treatment of TAK-925 group and the placebo group (each treatment of TAK-925 group - placebo group), the standard error and the two-sided 95% confidence intervals will be provided.

Property of Lakeda. For u

If there is a missing value of sleep latency in MWT at Day -1, it will be imputed by the predicted value of the same subject and the same session based on a model with sleep latency in MWT at Day -1 as a response, session as a fixed effect, and a subject as a random effect. After conducting imputation, the average sleep latency in MWT will be recalculated and the model analysis as above will be conducted as reference.



# Cohort C1~C2

Analysis Set: PD Set
Analytical

Method(s): The same analysis as section 7.9.2.1 "Cohort B1~B2" will be conducted.

7.9.2.2



7.9.2.3 CCI




7.9.2.4 CCI





7.9.2.5



7.9.2.6











7.9.2.8





7.10.1.2 <sup>CCI</sup>



7.10.1.3 <sup>CCI</sup>

CCI



#### **Safety Analysis** 7.11

In this study, safety will be evaluated as the primary endpoint.

#### 7.11.1 Adverse Events

7.11.1.1 Overview of Treatment-Emergent Adverse Events

#### Cohort A1~A3

Analysis Set: Safety Set

Analysis

Variable(s): **TEAE** 

applicable Terms of Use [Related, Not Related] Relationship to Study Drug Categories:

> [Mild, Moderate, Severe] Intensity

Analytical

The following summaries will be provided for each treatment group. Method(s):

(1) Overview of Treatment-Emergent Adverse Events

- 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
- 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 4) Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects)
- Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- 8) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

Property of Lakeda. For U.S. TEAEs will be counted according to the rules below. Percentages for each treatment group will be based on the number of subjects in the safety set. Number of subjects

• Summaries for 2) and 6)

• Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

Summaries other than 2), 3), and 6)

A subject with multiple • Summaries other than 2), 3), and 6)

## Number of events

For each summary, the total number of events will be calculated.

#### Cohort B1~B2

Analysis Set: Safety Set

Analytical

The same analysis as section 7.11.1.1 "Cohort A1~A3" will be performed Method(s):

for the Cohort B1~B2.

#### Cohort C1~C2

Analysis Set: Safety Set

Analytical

The same analysis as section 7.11.1.1 "Cohort A1~A3" will be performed Method(s):

for the Cohort C1~C2.

Safety Set Analysis Set:

Analytical

Method(s): The same analysis as section 7.11.1.1 "Cohort A1~A3" will be performed

for the Cohort A'1

7.11.1.2 Displays of Treatment-Emergent Adverse events

#### Cohort A1~A3

Analysis Set: Safety Set

Analysis

Variable(s): TEAE

Categories: Intensity [Mild, Moderate, Severe]

Time of Onset (day) [Day 1, Day 2, Day 3, Day 4, Day 5,

Day 6, Day 7, Day8 - Max]

Analytical

Probeith of Lakeda.

Method(s): The following summaries will be provided using frequency distribution for each treatment group.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (9) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (10) Treatment-Emergent Adverse Events Occurred during Infusion by System Organ Class and Preferred Term
- (11) Treatment-Emergent Adverse Events Occurred after Infusion by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below. Percentages for each treatment group will be based on the number of subjects in the safety analysis set.

#### Number of subjects

- Summary tables other than (5) and (6)
  A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT.
- Summary tables for (5) and (6)
   A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity.
- Summary table for (9)

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT.

When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

#### Cohort B1~B2

Analysis Set: Safety Set

Analytical\*

Method(s): The same analysis as section 7.11.1.2 "Cohort A1~A3" will be performed

for the Cohort B1~B2.

#### Cohort C1~C2

Analysis Set: Safety Set

Analytical

Method(s): The same analysis as section 7.11.1.2 "Cohort A1~A3" will be performed

for the Cohort C1~C2.

#### Cohort A'1

Analysis Set: Safety Set

Analysis

Variable(s): TEAE

Categories: Intensity [Mild, Moderate, Severe]

Analytical

Method(s): The following summaries will be provided using frequency distribution.

TEAEs will be coded using the MedDRA and will be summarized using

SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

# 7.11.1.3 Displays of Pretreatment Events

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): PTE

Analytical

Method(s): The following summaries will be provided using frequency distribution.

(erms of Use PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term
- (2) Serious Pretreatment Events by System Organ Class and Preferred

The frequency distribution will be provided according to the rules below.

## Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted icial use only and subject to only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

## 7.11.2 Clinical Laboratory Evaluations

### 7.11.2.1 Hematology and Serum Chemistry

#### Cohort A1~A3

Analysis Set: Safety Set

Analysis

Variable(s): Hematology

> **RBC** Hematocrit

Platelet **WBC** 

WBC Differentials (Neutrophils, Eosinophils, Basophils, Lymphocytes,

**MCHC MCV** 

Alkaline Phosphatase **ALT** 

Total Bilirubin Blood Urea Nitrogen

MCH
Serum Chemistry
Albumin
AST
Calc Chloride Creatinine Glucose Potassium

Sodium C-reactive Protein

**LDH** Magnesium Uric acid **Triglycerides** 

Predose, Day 4, Day 8, Day 15

(Data obtained at Day 1 will be used as the "Predose" visit)

Analytical

Method(s): The following summaries will be provided by treatment group.



#### Cohort B1~B2

Analysis Set: Safety Set

Analytical

The same analysis as section 7.11.2.1 "Cohort A1~A3" will be performed Method(s):

for the Cohort B1~B2.

#### Cohort C1~C2

Safety Set Analysis Set:

Analytical

Method(s): The same analysis as section 7.11.2.1 "Cohort A1~A3" will be performed

for the Cohort C1~C2.

Cohort A'1

Analysis Set: Safety Set

Visit: Predose, Day 2

(Data obtained at Day 1 will be used as the "Predose" visit)

Analytical

Method(s): The same analysis as section 7.11.2.1 "Cohort A1~A3" will be performed

for the Cohort A'1

#### 7.11.2.2 Urinalysis

#### Cohort A1~A3

Analysis Set: Safety Set

Analysis

Variable(s): Protein

, 4+]
, 2+, 3+]
[-, +-, +, 2+, 3+]
[5.0<= -<=7.5, 8.0<= -<=9.0]

7+-, +, 2+, 3+]
8, Day 15
1 will be used 2 Glucose Occult Blood

**Nitrite** 

Ketone Bodies

рН

Specific Gravity

Urobilinogen

Predose, Day 4, Day 8, Day 15 Visit:

(Data obtained at Day 1 will be used as the "Predose" visit)

Analytical

For Specific Gravity, summaries (1), (2) and (4) will be provided by Method(s):

treatment group.

For each variable other than Specific Gravity, summaries (3) and (4) will be

provided by treatment group.



#### Cohort B1~B2

Analysis Set: Safety Set

Analytical

Wie Leiths of Use The same analysis as section 7.11.2.2 "Cohort A1~A3" will be performed 3ct to the app Method(s):

for the Cohort B1~B2.

#### Cohort C1~C2

Analysis Set: Safety Set

Analytical

The same analysis as section 7.11.2.2 "Cohort A1~A3" will be performed use only and Method(s):

for the Cohort C1~C2.

#### Cohort A'1

Analysis Set: Safety Set

Visit: Predose, Day 2

(Data obtained at Day 1 will be used as the "Predose" visit)

Analytical

The same analysis as section 7.11.2.2 "Cohort A1~A3" will be performed Method(s):

for the Cohort A'1

#### 7.11.3











6 tobert



7.11.5 CCI

**Skobelg** 



7.11.6<sup>CCI</sup>





# 7.11.8 Other Observations Related to Safety

Not applicable.

#### 7.12 Interim Data Review

The dose level chosen for Cohorts in Part A, B, C after the first cohort in each group and whether to proceed to next cohort or stop the part may be evaluated by the sponsor's unblinded team composed of persons who do not have subject contact or involvement with execution of the protocol at the site, who will review unblinded data on safety, tolerability, available PK and PD results, and this dose may be higher, lower or the same than that used in the prior cohorts.

## 7.13 Changes in the Statistical Analysis Plan

From the SAP version 1.0, the following parts were updated. Cohort A3, C2 and A'1 were added in each section. Other main modified parts are as below.

Before the change

Cover

#### Prepared by:



Based on:

- - - ♦ Placebo (pooled Cohort B1 and B2)
  - Cohort C1
    - Placebo
    - TAK-925 TBD

## After the change

#### **Study Definitions**

- Treatment Group
  - Cohort A1~A3
    - ♦ Placebo (pooled Cohort A1, A2 and A3)
  - Cohort B1~B2
    - Placebo (pooled Cohort B1 and B2)

- Cohort C1<u>~C2</u>
  - ♦ Placebo
  - ♦ TAK-925 <u>44mg</u>, 112mg
- Cohort A'1

Reason for the change

The conducting cohorts and each dose level were determined.

Before the change

7.9.1.1 <sup>CCI</sup>



After the change



Property





Before the change

7.9.2.1 Average Sleep Latency in MWT/Sleep Latency in Each Session in MWT Cohort B1~B2

Analytical

The following summaries will be provided. Property of Takeda Method(s):

(1) For the average sleep latency in MWT, descriptive statistics for the changes from baseline and will be provided by visit by treatment group. The effect of TAK-925 will be evaluated with a linear mixed effects model. The response variable in the model will be the observed value of the average sleep latency in the MWT. The model will include treatment (each treatment of TAK-925 and placebo), day (as a categorical variable), the treatment-by-day as fixed effects, baseline average sleep latency in the MWT as a covariate, and subjects as a random effect. Least square (LS) means, the standard errors, and the two-sided 95% confidence intervals

will be provided for each treatment group. For each day, the difference in the LS means between each treatment of TAK-925 and the placebo (each treatment of TAK-925 - the placebo), the standard error of the difference and the two-sided confidence intervals will be provided.

The differences in the LS means between each treatment of TAK-925 group and the placebo group (each treatment of TAK-925 group - placebo group), the standard error and the two-sided 95% confidence intervals will be provided.

CCI

Property of Takeda. For no



7.9.2.1 Average Sleep Latency in MWT/Sleep Latency in Each Session in MWT/Cohort B1~B2

Analytical

Method(s): The following summaries will be provided.

(1) For the average sleep latent.

(1) For the average sleep latency in MWT, descriptive statistics for the , changes from baseline and will be provided by visit by treatment group. The effect of TAK-925 will be evaluated with a linear mixed effects model. The response variable in the model will be the change from baseline in the average sleep latency in the MWT. The model will include treatment (each average sleep latency in general variable variable variab treatment of TAK-925 and placebo), day (as a categorical variable), the treatment-by-day as fixed effects, baseline average sleep latency in the MWT as a covariate, and subjects as a random effect. Least square (LS) means, the standard errors, and the two-sided 95% confidence intervals will be provided for each treatment group. For each day, the difference in the LS means between each treatment of TAK-925 and the placebo

between each treatment of TAK-925 group and the placebo group (each



reference.



## Reason for the change

The response variable for model analysis was changed for better assessment. Because missing value was occurred at Day -1 of MWT value, the analysis using imputation method was added for reference.

## Before the change



After the change

7.9.2.2 <sup>CCI</sup>



TAK-925-1003

Reason for the change



To meet another department request.

Before the change

7.9.2.5



Reason for the change

Error correction.

Before the change

7.9.2.6

After the change

7.9.2.6 To meet another department request.

Before the change
7.9.2.7



After the change

7.9.2.7 <sup>CCI</sup>

Property





Error correction and adding another analysis variable and another analysis due to other department request.

Before the change
7.10.1

7.10.1

7.10.1.1 CCI





Before the change

Error correction and to clarify the description.

7.10.1 <sup>CCI</sup>

7.10.1.2 <sup>CCI</sup>



After the change

7.10.1 CCI

7.10.1.2 CC



Reason for the change

Error correction and to clarify the description.

Before the change

7.11.2.2 Urinalysis

Cohort A1~A2

Analysis

Variable(s): Protein [-, +-, +, 2+, 3+]

Glucose [-, +, 2+, 3+, 4+] Occult Blood [-, +-, +, 2+, 3+]

Nitrite [-, +]

Ketone Bodies [-, +-, +, 2+, 3+]

pH [5.0<= - <=7.5, 8.0<= - <=9.0]

Specific Gravity

Urobilinogen [+-, +, 2+, 3+]

Microscopy

RBC [below 1/HPF, 1-4/HPF, 5-9/HPF, 10-19/HPF,

20-29/HPF, 30-49/HPF, 50-99/HPF, above or equal to

100/HPF]

WBC [below 1/HPF, 1-4/HPF, 5-9/HPF, 10-19/HPF,

20-29/HPF, 30-49/HPF, 50-99/HPF, above or equal to

100/HPF]

Casts [below 1/HPF, 1-4/HPF, 5-9/HPF, 10-19/HPF,

20-29/HPF, 30-49/HPF, 50-99/HPF, above or equal to

100/HPF1

Visit: Predose, Day 4, Day 8, Day 15

(Data obtained at Day 1 will be used as the "Predose" visit)

Analytical

Method(s): For Specific Gravity, summaries (1), (2) and (4) will be provided by

treatment group.

For Microscopy (Erythrocytes (RBC), Leukocytes (WBC), Squamous

Cells), summaries (3) will be provided by treatment group.

For each variable other than Specific Gravity and Microscopy, summaries

(3) and (4) will be provided by treatment group.

After the change

7.11.2.2 Urinalysis

C

### Cohort A1~A3

### Analysis

[-, +-, +, 2+, 3+] Variable(s): Protein

> [-, +, 2+, 3+, 4+]Glucose [-, +-, +, 2+, 3+] Occult Blood

[-, +] **Nitrite** 

Ketone Bodies [-, +-, +, 2+, 3+]

[5.0<= - <= 7.5, 8.0<= - <= 9.0] pH

Specific Gravity

[+-, +, 2+, 3+]Urobilinogen

Visit: Predose, Day 4, Day 8, Day 15

se" vi (Data obtained at Day 1 will be used as the "Predose" visit)

Analytical

For Specific Gravity, summaries (1), (2) and (4) will be provided by Method(s):

treatment group.

For each variable other than Specific Gravity, summaries (3) and (4) will be

provided by treatment group. Mercial USE

Reason for the change

Error correction.

#### Before the change

7.11.3.1



Reason for the change

Error correction and to clarify the description.

Sie Terms of Use Before the change 7.11.4 After the change 7.11.4 mercial use only Reason for the change Error correction. Before the change 7.11.5

After the change

7.11.5



Reason for the change

asis for chat as for chat and subject to mondommercial use only and subject to mondommercial use of the To make the definitions more appropriate and the analysis for change from time-matched day 1 to day 7 was added

